CLINICAL TRIAL: NCT03656614
Title: Dose Finding Study for Reversal of Vecuronium-induced Neuromuscular Blockade at Train-of-four Ratio 0.3 With Sugammadex and Neostigmine
Brief Title: Reversal of Residual Neuromuscular Blockade at Train-of-four Ratio 0.3 With Sugammadex and Neostigmine
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: Reversal Neuromuscular Block
Record Dates: First submitted 2018-07-10; First posted 2018-09-04 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Neuromuscular Blockade
Keywords: sugammadex neostigmine
MeSH Terms: interventions — Sugammadex; Neostigmine; Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (11):
- sugammadex 0.125: Sugammadex group: sugammadex 0.125 mg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Sugammadex
- Sugammadex 0.25: Sugammadex group: sugammadex 0.25 mg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Sugammadex
- Sugammadex 0.5: Sugammadex group: sugammadex 0.5 mg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Sugammadex
- Sugammadex 1.0: Sugammadex group: sugammadex 1.0 mg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Sugammadex
- Sugammadex 2.0: Sugammadex group: sugammadex 2.0 mg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Sugammadex
- Neostigmine 10: Neostigmine group: neostigmine 10 µg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Neostigmine
- Neostigmine 25: Neostigmine group: neostigmine 25 µg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Neostigmine
- Neostigmine 40: Neostigmine group: neostigmine 40 µg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Neostigmine
- Neostigmine 55: Neostigmine group: neostigmine 55 µg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Neostigmine
- Neostigmine 70: Neostigmine group: neostigmine 70 µg/kg IV once at the reappearance of TOF 0.3
  Interventions: Drug: Neostigmine
- Placebo: Placebo group: Saline 0.9% IV once at the reappearance of TOF 0.3
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Sugammadex — At the end of surgical procedure at a depth of neuromuscular blockade at the reappearance of train-of-four 0.3, single intravenous injection of either :
  Sugammadex 0.125 mg/kg (sugammadex 0.125) Sugammadex 0.25 mg/kg (sugammadex 0.25) Sugammadex 0.5 mg/kg (sugammadex 0.5) Sugammadex 1.0 mg/kg (sugammadex 1.0) Sugammadex 2.0 mg/kg (sugammadex 2.0)
  Other Names: Bridion; Org 25969
  Groups: Sugammadex 0.25; Sugammadex 0.5; Sugammadex 1.0; Sugammadex 2.0; sugammadex 0.125
Drug: Neostigmine — At the end of surgical procedure at a depth of neuromuscular blockade at the reappearance of train-of-four 0.3, single intravenous injection of either :
  Neostigmine 10 µg/kg (Neostigmine 10) Neostigmine 25 µg/kg (Neostigmine 25) Neostigmine 40 µg/kg (Neostigmine 40) Neostigmine 55 µg/kg (Neostigmine 55) Neostigmine 70 µg/kg (Neostigmine 70)
  Atropine will be administered with Neostigmine at a half dose of Neostigmine administered through an intravenous line with brisk flow.
  Other Names: Prostigmin
  Groups: Neostigmine 10; Neostigmine 25; Neostigmine 40; Neostigmine 55; Neostigmine 70
Drug: Saline 0.9% — At the end of surgical procedure at a depth of neuromuscular blockade at the reappearance of train-of-four 0.3, single intravenous injection of saline 0.9%.
  Other Names: Placebo
  Groups: Placebo

SUMMARY:
The aim of this study is to estimate the optimal dose of sugammadex and neostigmine reversal of a vecuronium-induced residual neuromuscular block at train-of-four ratio 0.3.

DETAILED DESCRIPTION:
Sugammadex is a modified γ-cyclodextrin compound that reverses the neuromuscular blockade produced by steroidal nondepolarizing muscle relaxants such as rocuronium,vecuronium and pipecuronium by encapsulating them, making them unavailable to interact with the nicotinic acetylcholine receptors at the neuromuscular junction.However, residual neuromuscular blocks between reappearance of T4 and train-of-four ratio (TOFR)=0.5 are more frequent in clinical practice compared with profound or deep blocks and have not been investigated for sugammadex previously.

Unlike neostigmine, sugammadex is efficacious in reversing profound (no responses to either train-of-four (TOF) or posttetanic count stimulation) or deep (posttetanic count of 1 or 2) neuromuscular block (NMB) in doses of 16 and 4 mg/kg, respectively. However, shallow neuromuscular blocks are more frequent in clinical practice compared with profound or deep blocks and have not been investigated for sugammadex previously.

ELIGIBILITY:
Inclusion Criteria:

* 1 age of 18 to 65 yr,
* 2 body mass index 18.5 to 25.0 kg/m2,
* 3 American Society of Anesthesiologists physical status I to III
* 4 scheduled for elective surgery with an expected duration of at least 60min under general anesthesia with intubation of the trachea or laryngeal mask
* 5 patients having given informed consent to the study

Exclusion Criteria:

* 1 patients who had participated in another clinical trial within 1 month
* 2 Patients with suspected difficult airway, bronchial asthma, chronic obstructive pulmonary disease
* 3 known neuromuscular disease
* 4 suspected malignant hyperthermia
* 5 hepatic or renal dysfunction
* 6 glaucoma
* 7 allergy to the medication that used in this trial
* 8 taking medicaments that might influence the effect of NMB agents
* 9 pregnant, or breastfeeding state
* 10 taking medication known to alter the effect of neuromuscular blocking agents( toremifene .etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people scheduled for elective surgery
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Time to TOF 0.9 after the administration of reversal agent | the general anesthesia time 1 hour at least
  The time to achieve TOF (Train of Four stimulation) ratio to 0.9 following the investigational drug or placebo administration.

SECONDARY OUTCOMES:
incidence of reparalysis | approximately 1 hour
  Determining whether patients receiving reversal agent will have a train-to-four ratio <0.8 during total recovery time (from TOF reach 0.9 first time to post-anaesthesia care unit (PACU) departure)
incidence of adverse event | the general anesthesia and recovery time 2 hours at least
  Documenting whether patients will have some adverse events(such as hypoxia bradycardia nausea and vomiting) from anesthesia commence to PACU departure.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Pongracz A, Szatmari S, Nemes R, Fulesdi B, Tassonyi E. Reversal of neuromuscular blockade with sugammadex at the reappearance of four twitches to train-of-four stimulation. Anesthesiology. 2013 Jul;119(1):36-42. doi: 10.1097/ALN.0b013e318297ce95. PMID 23665915
- [Background] Schaller SJ, Fink H, Ulm K, Blobner M. Sugammadex and neostigmine dose-finding study for reversal of shallow residual neuromuscular block. Anesthesiology. 2010 Nov;113(5):1054-60. doi: 10.1097/ALN.0b013e3181f4182a. PMID 20885293
- [Background] Kaufhold N, Schaller SJ, Stauble CG, Baumuller E, Ulm K, Blobner M, Fink H. Sugammadex and neostigmine dose-finding study for reversal of residual neuromuscular block at a train-of-four ratio of 0.2 (SUNDRO20)dagger, Br J Anaesth. 2016 Feb;116(2):233-40. doi: 10.1093/bja/aev437. PMID 26787792
- [Derived] He J, He H, Li X, Sun M, Lai Z, Xu B. Required dose of sugammadex or neostigmine for reversal of vecuronium-induced shallow residual neuromuscular block at a train-of-four ratio of 0.3. Clin Transl Sci. 2022 Jan;15(1):234-243. doi: 10.1111/cts.13143. Epub 2021 Nov 2. PMID 34435439